CLINICAL TRIAL: NCT05482022
Title: Speaking Valve Influence on Breathing, Swallowing and Vocal Functions in Patients With Tracheostomy.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loewenstein Hospital (Other)
Responsible Party: Principal Investigator, elena eidinov, Head of Intensive Care for Consciousness Rehabilitation Department, Loewenstein Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0027-21-LOE
Record Dates: First submitted 2022-07-25; First posted 2022-08-01 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Tracheostomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- speaking valve (Experimental): Respiratory physical therapy treatments conducted using a speaking valve for 2 weeks (at least 8 treatments).
  Interventions: Device: Shiley™ phonate speaking valve
- control (Other): Respiratory physical therapy treatments conducted without using a speaking valve .
  Interventions: Other: control

INTERVENTIONS:
Device: Shiley™ phonate speaking valve — The device connects to the tracheostomy tube. Usually used to aid vocalization.
  Other Names: speaking valve
  Arms: speaking valve
Other: control — no intervention
  Arms: control

SUMMARY:
Speaking valve seems to have a beneficial influence on breathing and secretion management in certain patients with tracheostomy.

The investigators plan to use a speaking valve during respiratory physical therapy sessions in participants with disturbances of consciousness, who have a tracheostomy, with no need of a mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* brain injury (traumatic/non-traumatic).
* tracheostomy.
* unresponsive wakefulness syndrome or minimally conscious state.
* fiber optic examination as follows: good mobilization of the vocal cords. No airway granulation, MarianJoy scale score: 1-3.
* the legal guardian speaks Hebrew.

Exclusion Criteria:

* airway stenosis / inflammation.
* oxygen saturation <90%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
change from baseline oxygen saturation | 15 minutes
  at physical therapy sessions
change from baseline breathing rate | 15 minutes
  at physical therapy sessions

SECONDARY OUTCOMES:
rate of swallowing | 15 minutes
  during a physical therapy session
percentage of participants presenting vocalization | 2 weeks
  occurrence of vocalization at the respiratory physical therapy sessions.
cough rate | 2 weeks
  the ratio of respiratory physical therapy sessions eliciting cough.
percentage of patients weaned from tracheostomy | through study completion, an average of 6 months.
  whether or not decannulation was successfully performed during rehabilitation.

OTHER OUTCOMES:
number of desaturation events | 2 weeks
  oxygen levels decrease below 90% or by 3% from baseline during respiratory physical therapy sessions.
number of respiratory physical therapy sessions | 2 weeks
  the number of respiratory physical therapy sessions given to a participant

CONTACTS AND LOCATIONS:
Locations (1):
- Loewenstein Rehabilitation Hospital, Raanana, Israel

IPD SHARING:
Plan to Share IPD: No